CLINICAL TRIAL: NCT06195501
Title: Transoesophageal Echocardiography - Dysphagia Risk in Acute Stroke- TEDRAS 2 - Follow Up
Brief Title: Dysphagia After Transesophageal Echocardiography in Acute Stroke - Follow Up Trial
Acronym: TEDRAS2
Status: Recruiting | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Samra Hamzic, Prinicipal Investigator, University of Giessen
Other Study IDs: TEDRAS2
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Ischemic Stroke, Acute; Dysphagia Following Cerebrovascular Accident
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute ischemic stroke: Patients with acute ischemic stroke and an indication for a transesophageal ecocardiography
  Interventions: Diagnostic Test: Flexible Endoscopic Evaluation of Swallowing (FEES) ; Transesophageal Ecocardiography (TEE)

INTERVENTIONS:
Diagnostic Test: Flexible Endoscopic Evaluation of Swallowing (FEES) ; Transesophageal Ecocardiography (TEE) — Flexible Endoscopic Evaluation of Swallowing (FEES):
  FEES is performed for analysis of swallowing ability according to the same methodology as in the initial trial: one day before a TEE and max. 4 hours after TEE. Before the FEES anticongestive nose drops are applied and the nostrils are anaesthetized by applying a lidocaine gel via cotton sticks. During the FEES examination the participants sit upright and are asked to swallow various consistencies: FEES is aborted in case of aspiration of any of the consistencies during the examination.
  Transesophageal Ecocardiography (TEE):
  For the TEE anesthesia is applied via intravenous injection of propofol or a combined anesthesia, through intravenous application of propofol and local anesthesia, using lidocaine spray. All patients undergoing a TEE are sober before and at least two to four hours after TEE.

SUMMARY:
The aim of the prospective observational TEDRAS - Follow-up Trial is to investigate the limitations of the initial TEDRAS - Trial in patients with acute Dysphagia is a common consequence from ischemic stroke and it correlates with an increased risk of pulmonary complications such as aspiration pneumonia and an increased mortality risk.

TEDRAS-Trial (Transesophageal Echocardiography: Dysphagia Risk in the Acute Phase After Stroke; ClinTrial.gov identifier NCT04302883) was the first randomized and controlled trial to address the question of the extent to which TEE increases dysphagia risk in acute stroke patients. The results of the study confirmed the hypothesis that dysphagia severity worsens after TEE in the intervention group.

The aim of the prospective observational TEDRAS - Follow-up Trial is to investigate the limitations of the initial TEDRAS - Trial in patients with acute ischemic stroke.

DETAILED DESCRIPTION:
Dysphagia is a common consequence from ischemic stroke and it correlates with an increased risk of pulmonary complications such as aspiration pneumonia and an increased mortality risk.

Early detection of dysphagia increases the overall outcome, reduces the mortality risk, the risk of aspiration pneumonia, malnutrition as well as the length of hospitalization and the overall costs of treatment.

In German stroke units within 24 hours of admission stroke patients undergo a clinical swallowing screening and the flexible endoscopic evaluation of swallowing (FEES), if necessary. FEES allows for a valid assessment of swallowing and description of dysphagia symptoms via standardized scores as the Secretion Severity Sating Scale (SSRS), the Penetration-Aspirations-Scale (PAS), the Yale Pharyngeal Residue Severity Scale (YSPRSS) and the Functional Oral Intake Scale (FOIS-G).

Transesophageal echocardiography (TEE) is conducted within the first few days after stroke as a routine examination to detect whether a cardiac disorder was the cause of stroke. The implementation of a TEE during cardiac surgery has a significant correlation with occurrences of postoperative dysphagia in patients after cardiac surgery [1].

TEDRAS-Trial (Transesophageal Echocardiography: Dysphagia Risk in the Acute Phase After Stroke; ClinTrial.gov identifier NCT04302883) [2] was the first randomized and controlled trial to address the question of the extent to which TEE increases dysphagia risk in acute stroke patients. The results of the study confirmed the hypothesis that dysphagia severity worsens after TEE in the intervention group [2].

The aim of the prospective observational TEDRAS - Follow-up Trial is to investigate the limitations of the initial TEDRAS - Trial in patients with acute ischemic stroke.

In particular, the following parameters will be examined:

1. The influence of the type and route (intravenous vs. oral) of anesthesia administered during TEE on swallowing in all cohorts studied.
2. The correlation between the duration of TEE and the degree of deterioration in FOIS-G after TEE.
3. The interrater reliability for the FEES.
4. Definition of typical dysphagia symptoms after TEE.

ELIGIBILITY:
Inclusion Criteria:

* Acute cerebral infarction detected by cMRI or cCT
* Indication for TEE
* Neurological deficits
* Written informed consent

Exclusion Criteria:

* Cerebral hemorrhage
* Contraindications to FEES (lack of alertness as well as lack of compliance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke and indication for TEE
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Penetration-Aspiration-Score (PAS) | Immediately after the intervention
  Penetration-Aspiration-Score, minimum value 1, maximum value 8; higher scores mean worse outcome
Functional Oral Intake Scale-German (FOIS-G) | Immediately after the intervention
  Functional Oral Intake Scale - German Version; minimum value 1, maximum value 7; higher scores mean better outcome
Yale Scale (YS) | Immediately after the intervention
  Yale Pharyngeal Residue Severity Rating Scale; minimum value 1, maximum value 5; higher scores mean worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Samra Hamzic, Dr, Principal Investigator — University Hospital Giessen and Marburg, Campus Giessen
Locations (1):
- University Hospital Giessen and Marburg, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hamzic S, Braun T, Butz M, Khilan H, Weber S, Yeniguen M, Gerriets T, Schramm P, Juenemann M. Transesophageal Echocardiography - Dysphagia Risk in Acute Stroke (TEDRAS): a prospective, blind, randomized and controlled clinical trial. Eur J Neurol. 2021 Jan;28(1):172-181. doi: 10.1111/ene.14516. Epub 2020 Oct 10. PMID 32897605
- [Derived] Hamzic S, Juenemann M, Braun T, Piayda K, Bauer P, Sossalla S, Gerriets T, Khilan H, Butz M, Schramm P, Omar OA. TEDRAS II - transesophageal echocardiography as dysphagia risk in the acute phase of stroke-protocol for a prospective pilot observational trial. Trials. 2025 Oct 27;26(1):445. doi: 10.1186/s13063-025-09065-5. PMID 41146308
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/32897605/